CLINICAL TRIAL: NCT00243256
Title: Treatment of Obesity With Vitamin D (40.000 IE Per Week for 1 Year)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tromso (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSEMDT-2005-2
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol

SUMMARY:
The purpose of the study is to evaluate if supplementation with vitamin D in doses of 20.000IU per week and 40.000 IU per week will result in weight loss in obese subjects as compared to placebo during 1 year.

DETAILED DESCRIPTION:
We will include 450 obese subjects that will be devided in 3 groups: 40.000IU cholecalciferol per week, 20.000 IU cholecalciferol per week, and placebo. All subjects will be given 500 mg calcium per day. There will be visits every tird month. In addition to weight reduction, we will also evaluate the calcium metabolism (blood test and urin samples), insulin sensitivity, muscle strenght, blood pressure and depression.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 - 40
* serum calcium < 2.55 mmol/L

Exclusion Criteria:

* serious diseases
* reduced kidney function
* renal stone disease
* using psychopharmaca
* using drugs for weight reduction

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2005-11; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Body Weight
Body composition
Measures of calcium metabolism
Insulin sensitivity
Muscle strength
Depression score
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromsø, Tromsø, Norway
Locations (1):
- Clinical Research Unit, University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Jorde R, Sneve M, Torjesen PA, Figenschau Y, Hansen JB, Grimnes G. No significant effect on bone mineral density by high doses of vitamin D3 given to overweight subjects for one year. Nutr J. 2010 Jan 7;9:1. doi: 10.1186/1475-2891-9-1. PMID 20056003